CLINICAL TRIAL: NCT07207837
Title: Effect of Stress Ball Use on Pain, Sleep Quality and Physiological Parameters in Critically Ill: Randomized Controlled Trial
Brief Title: Effect of Stress Ball Use on Pain, Sleep Quality and Physiological Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Yeşim Yaman Aktaş, Professor, Giresun University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: yesim.yaman
Record Dates: First submitted 2025-09-17; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Critically Ill Patients Admitted in ICU
Keywords: critically ill patients; pain; sleep quality; stress ball
MeSH Terms: conditions — Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): In the experimental group, after the VAS assessment at 22.00 pm on the second day, a stress ball was applied between 22:30-22:45 pm before going to sleep at night. Patients were given a round, silicone, medium-sized and medium-hard stress ball, and were asked to squeeze it for a total of 15 minutes (counting from one to five and squeezing 2 times in each application), allowing them to rest from time to time as they wished. After the stress ball application, physiological parameters were measured every two hours from 01.00 at night. In the experimental group, all data collection procedures were completed by re-evaluating the VAS and RCQ at 07.00 in the morning. In this study, physiological parameters in both groups were collected in 4 periods during the day (01.00-05.00 at night, 07.00-11.00 in the morning, 13.00-17.00 at noon, 19.00-23.00 in the evening) and the averages of the measurement values obtained in each period were used in the analysis.
  Interventions: Other: Stress Ball Use
- Control group (No Intervention): In patients admitted to the ICU, diagnostic forms were filled out on the first night and physiological parameters (blood pressure, pulse rate, respiratory rate, body temperature) of both groups were monitored within the scope of standard care every two hours starting from 01.00 h and VAS and RCUQ were applied to all participants at 07.00 h in the morning. On the second day, only standard care was provided to the control group, VAS was recorded at 22.00 p.m., physiological parameters were recorded every two hours from 01.00 a.m., and VAS and RCQ were applied again at 07.00 a.m.

INTERVENTIONS:
Other: Stress Ball Use — The stress ball suppresses most of the nerves and muscles around the wrist and hand, which are directly connected to the brain, and stimulates the nerves and muscles. This mechanism reduces the release of stress hormones and regulates blood pressure by providing relaxation and relaxation (Dinis & Sousa, 2023; Soltani et al., 2023). Stress ball, which is easy to apply, inexpensive, has no side effects on the patient, and is an effective method in physical and emotional recovery, is an intervention that can be preferred in nursing practices (Gezginci, Iyigun, Kibar, & Bedir, 2018; Kasar, Erzincanli, & Akbas, 2020). Stress ball application is effective on pain, anxiety and vital signs in different patient groups (Genç, Korkmaz, & Akkurt, 2022; Gezginci, Iyigun, Kibar, & Bedir, 2018; Karatas & Gezginci, 2023), but no randomised controlled study has been found in which stress ball application was performed in intensive care patients.
  Arms: experimental group

SUMMARY:
Environmental stressors, pain and sleep disorders are common in intensive care patients and non-pharmacological approaches can be effective in the management of these factors. This study will be conducted to investigate the effect of stress ball use on pain, sleep quality and physiologic parameters in critically ill patients. The study is a randomised controlled study. In this study, Patient Information Form, Glasgow Coma Scale and Ramsey Sedation Scale, Visual Analogue Scale (VAS), Richard-Campbell Sleep Scale (RCS) will be used to collect data. Patients who were admitted to the intensive care unit and met the research criteria will be assigned to the experimental or control group and their verbal and written consents were obtained. Intensive care nurses can contribute to improving the sleep quality of patients, reducing pain and improving some physiological parameters with stress ball application.

DETAILED DESCRIPTION:
Intensive care units (ICU) are environments where critically ill patients are treated and require advanced medical intervention . Critically ill patients in ICU are monitored from the time of admission and their physiological parameters such as blood pressure, heart rate, respiratory rate, oxygen saturation are closely monitored. In addition to the existing diseases of patients in intensive care units, the presence of many technological devices such as haemodynamic monitoring required for follow-up and treatment and the complex nature of intensive care services often cause patients to experience pain .

More than 50% of intensive care patients experience pain due to surgical intervention, invasive procedures and morbidity. It is reported that patients experience 30% pain during rest and 50% pain during routine nursing practices such as endotracheal aspiration, deep breathing and coughing exercises, positioning, wound care, and catheter placement due to health problems. However, it is seen that pain management is generally inadequate and this situation affects the physical and psychological recovery processes of patients. The whole organism can be affected by pain, and accordingly, physiological and behavioural symptoms may occur in individuals experiencing pain. After the neuroendocrine response to pain, heart rate, cardiac output, myocardial oxygen consumption and peripheral vascular resistance increase as physiological symptoms.

In intensive care units where critically ill patients are followed up, changes in physiological parameters due to pain and other factors can be life-threatening. Defining pain, evaluating physiological parameter changes, and reducing or eliminating pain with the right nursing interventions is an important responsibility for nurses in specialised units such as intensive care. However, due to the critical condition of patients in the intensive care unit, patients may not be able to express pain subjectively and nurses may be inadequate in pain assessment. Generally, pain management is performed according to the physician's order, and appropriate nursing diagnoses cannot be made due to inadequate knowledge of nurses about pain. Inadequate pain treatment causes sleep deprivation, which is frequently seen in intensive care patients.

In intensive care units, many factors other than pain (e.g., constantly bright environment in intensive care, medical devices and sounds made by medical devices, IV drug treatments, lack of attention to privacy, too cold or hot environment and mechanical ventilation, etc.) can cause sleep problems by causing excessive stimulation. Sleep is a critical part of the healing process; however, ICU patients often do not get enough sleep. In addition to its negative effects on the immune system, sleep deprivation may also impair the general well-being of patients and prolong their recovery time. Therefore, improving sleep quality in ICU can accelerate the treatment process of patients and increase their general well-being. Intervening in environmental factors, for example, reducing the lights in the environment and muting or switching off the sound of vital medical devices, carries a great risk. For this reason, it may be easier to change patients' perception of the environment rather than changing the environment. It is especially recommended to use non-pharmacological methods to reduce the perception of the environment.

Although pharmacological treatment options are available for the management of these psychological and physiological burdens in intensive care patients, in recent years, non-pharmacological methods have increasingly found a place in the care of intensive care patients. One of these methods is the use of a stress ball. The stress ball, which is a low-cost and easily applicable method, can provide physical relief to patients. The stress ball suppresses most of the nerves and muscles around the wrist and hand, which are directly connected to the brain, and stimulates the nerves and muscles. This mechanism reduces the release of stress hormones and regulates blood pressure by providing relaxation and relaxation. Stress ball, which is easy to apply, inexpensive, has no side effects on the patient, and is an effective method in physical and emotional recovery, is an intervention that can be preferred in nursing practices. Stress ball application is effective on pain, anxiety and vital signs in different patient groups, but no randomised controlled study has been found in which stress ball application was performed in intensive care patients. In this study, it was aimed to examine the effect of stress ball use on pain, sleep quality and physiological parameters in intensive care patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agreed to participate in the study, who were older than 18 years of age, who could speak and understand Turkish, who had been treated in the ICU for at least 48 hours, who had a score of 15 on the Glasgow Coma Scale and a score of 2 on the Ramsey Sedation Scale, who were extubated, who had not received intravenous sedation and anaesthetic drugs for the last 12 hours, who could communicate meaningfully, and who did not have a physical disability in squeezing the stress ball were included in the study.

Exclusion Criteria:

* Patients using antihypertensive, beta blockers and similar drugs, experiencing situations that would cause them to leave the study (death, transfer to another unit, discharge or unwillingness to continue the study, etc.), receiving inotropic treatment (dopamine, steradine and others), patients with hearing and vision problems, patients treated with a diagnosis of sleep disorder, patients with a diagnosis of depression and anxiety disorder and treated with this diagnosis, patients with analgesic treatment in routine treatment were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Effect of Stress Ball Use on Pain in Critically Ill | 2 months
  This scale, which is used to determine the intensity of the pain felt, aims for the patient to express their pain in numbers. It was developed to convert a subjective value that cannot be measured numerically into a numerical value (Eren & Öztürk, 2021). It is usually 10 cm long and is a line starting with the absence of pain and progressing to the level of unbearable pain. In this study, a scale ranging from 0 to 100 was used and the patient was asked to indicate the number at which the pain reached. In the scale, the absence of pain was evaluated with 0 points and the most severe pain scoring was evaluated as 100 points.

SECONDARY OUTCOMES:
Effect of Stress Ball Use on Sleep Quality in Critically Ill Patients | 2 months
  Richard-Campbell Sleep Questionnaire (RCSQ): It was developed by Richards in 1987 and adapted into Turkish by Karaman Özlü and Özer. This scale consists of 6 items evaluating sleep quality, depth of sleep at night, frequency of awakening, ambient sound level, time of staying awake and time to fall asleep. Each item is evaluated on a scale of 0-100. A score between "0-25" indicates very poor sleep and a score between "76-100" indicates very good sleep. The Cronbach Alpha value of the Turkish form of the scale was found to be 0.91 (Karaman Özlü & Özer, 2015)

CONTACTS AND LOCATIONS:
Overall Officials: Yeşim Yaman Aktaş, Professor, Principal Investigator — Giresun University
Locations (1):
- Giresun University Health Sciences Faculty, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No